CLINICAL TRIAL: NCT00974038
Title: Cognitive Behavior Therapy for Adolescents With Bulimia Nervosa
Brief Title: Cognitive Behavior Therapy for Adolescents With Bulimia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4819
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Bulimia Nervosa
Keywords: Bulimia Nervosa, EDNOS, Adolescents
MeSH Terms: conditions — Bulimia Nervosa | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBT, SP (Experimental): cognitive behavioral therapy, supportive psychotherapy
  Interventions: Behavioral: psychotherapy

INTERVENTIONS:
Behavioral: psychotherapy — 1) cognitive-behavioral therapy or 2) supportive psychotherapy

SUMMARY:
We are interested in studying two different psychological treatments for eating disorders for adolescents (ages 12-18). The study is designed to help adolescents who are having problems with binge eating and/or purging. The treatment consists of 14 sessions of approximately one-hour each over about three months.

DETAILED DESCRIPTION:
Interested adolescents will have a phone screen and then come in for an in-person psychiatric evaluation. If eligible and interested, they will be randomly assigned to 4 months of outpatient treatment (free of charge) that is either 1) cognitive-behavioral therapy or 2) supportive psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Current or prior DSM IV diagnosis of Bulimia Nervosa or Sub-threshold Bulimia Nervosa (those who meet all DSM-IV criteria for BN, but engage in subjective binge-eating episodes and binge/purge at a frequency of at least once per week for 3 months, whereas meeting full DSM-IV criteria for BN requires binge eating and purging twice per week for 3 months)
* Major Depression

Exclusion Criteria:

* Diagnosis of bipolar disorder, current psychosis, drug or alcohol abuse in past 3 months, acute suicidal risk, major depression producing significant functional impairment, significant medical illness, weight outside of normal weight range.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2006-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Binge-eating a purging (EDE scores) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Sysko, Ph.D., Study Director — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States